CLINICAL TRIAL: NCT02211651
Title: Maternal Adipose Tissue and Placental Dysfunction Programs the Fetus for Type 2 Diabetes (PlacentA-DM)
Acronym: PlacentA-DM
Status: Completed | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: Sanford-Burnham Medical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TRIMDFH 499458; 499458 (Other: Florida Hospital IRB)
Record Dates: First submitted 2014-05-16; First posted 2014-08-07 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: adipose tissue; placenta; pregnancy; umbilical cord
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood Adipose tissue Placental tissue Umbilical Cord tissue Umbilical Cord blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- ObeseDYS: Obese subjects with dysfunctional vascularization and inflammation of placenta.
- ObeseNL: Obese subjects with normal vascularization and inflammation of placenta
- LeanNL: Lean subjects with normal vascularization and inflammation of placenta.

SUMMARY:
The purpose of this study is to discover the characteristics of pregnant women which increases risk for their babies to develop diabetes, later on in life.

DETAILED DESCRIPTION:
Obesity has been recently diagnosed in a younger population and currently in the United States more than two thirds of women of childbearing age are overweight or obese. These women will have children at high risk for developing obesity and Type 2 diabetes (T2DM). There is an acute need for preventing these complications in children so that we can break the cycle of obesity and T2DM. Numerous interventions have attempted but failed to improve outcomes in obese pregnancies by weight loss. Clinicians do not currently have specific recommendation for identifying the obese mothers and risk and for the prevention of infant's complication in healthy obese pregnancies.

The global objective of this study is to identify the relevant maternal phenotype at risk and the mechanism(s) of fetal environment predisposing the offspring for T2DM. This will enhance T2DM early screening and prevention.

The global hypothesis is that dysfunctional adipose tissue secretes angiostatic and pro-inflammatory factors that lead to the formation of a dysfunctional placenta, which through a hypoxic and inflamed environment alters the epigenome to program the fetus for T2DM.

ELIGIBILITY:
Pregnant women Inclusion Criteria:

* Pregnant women undergoing planned cesarean section at 39 weeks of gestation due to: a) elective cesarean section; b) breach presentation c) repeat cesarean section (the rationale for choosing these women is to select only women that have no other risk factors or complications during pregnancy that might affect the outcome)
* Age between 18 and 40 years old
* Pre-pregnancy BMI between 20 and 25 kg/m2 (lean) and >30 kg/m2 (obese)
* Singleton pregnancies
* Allowing their neonates to participate in the trial

Pregnant women Exclusion Criteria:

* Taking any medication except pre-natal vitamins and medication to treat normal symptoms of pregnancy like: constipation, nausea, vomiting, gastric reflux, insomnia and pain.
* Type 1 diabetes, type 2 diabetes or gestational diabetes; chronic or gestational hypertension
* Pre-eclampsia, eclampsia during this pregnancy
* Liver, kidney, thyroid disease, cancer
* Smoking or using illegal drugs or alcohol during this pregnancy
* Fetal umbilical blood and/or placenta are collected for another reason, i.e. parents decide on cord blood storage

Neonate Inclusion criteria:

- Live neonates born to the study participating mothers

Neonate exclusion criteria:

- Neonate distress as to require admission to the Neonatal Intensive Care Unit.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Vulnerable populations- Pregnant Women, Fetuses and Neonates
  Propose to study pregnant women in order to determine the relevant phenotype with offspring at risk for obesity and T2DM.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Quantity of Blood Vessels and Capillaries | Visit 3, at 39 weeks
  Measurements will be immunohistochemistry and measured from placental tissue. Neonate's anthropometrics and sex will be recorded within 48 hours of the delivery by the Pediatrician and will last approximately 15 minutes.
Quantity of macrophages | Visit 3 at 39 weeks + 1 day
  Measured by immunohistochemistry, flow cytometry (FACS) of placental tissue

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Smith, MD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

REFERENCES:
- [Background] Ling C, Groop L. Epigenetics: a molecular link between environmental factors and type 2 diabetes. Diabetes. 2009 Dec;58(12):2718-25. doi: 10.2337/db09-1003. No abstract available. PMID 19940235
- [Background] Dabelea D, Crume T. Maternal environment and the transgenerational cycle of obesity and diabetes. Diabetes. 2011 Jul;60(7):1849-55. doi: 10.2337/db11-0400. No abstract available. PMID 21709280
- [Background] Sullivan EL, Smith MS, Grove KL. Perinatal exposure to high-fat diet programs energy balance, metabolism and behavior in adulthood. Neuroendocrinology. 2011;93(1):1-8. doi: 10.1159/000322038. Epub 2010 Nov 13. PMID 21079387
- [Background] Catalano PM, Farrell K, Thomas A, Huston-Presley L, Mencin P, de Mouzon SH, Amini SB. Perinatal risk factors for childhood obesity and metabolic dysregulation. Am J Clin Nutr. 2009 Nov;90(5):1303-13. doi: 10.3945/ajcn.2008.27416. Epub 2009 Sep 16. PMID 19759171
- [Background] Crume TL, Ogden L, Daniels S, Hamman RF, Norris JM, Dabelea D. The impact of in utero exposure to diabetes on childhood body mass index growth trajectories: the EPOCH study. J Pediatr. 2011 Jun;158(6):941-6. doi: 10.1016/j.jpeds.2010.12.007. Epub 2011 Jan 15. PMID 21238981
- [Background] Dabelea D, Mayer-Davis EJ, Lamichhane AP, D'Agostino RB Jr, Liese AD, Vehik KS, Narayan KM, Zeitler P, Hamman RF. Association of intrauterine exposure to maternal diabetes and obesity with type 2 diabetes in youth: the SEARCH Case-Control Study. Diabetes Care. 2008 Jul;31(7):1422-6. doi: 10.2337/dc07-2417. Epub 2008 Mar 28. PMID 18375420
- [Background] Catalano PM, Presley L, Minium J, Hauguel-de Mouzon S. Fetuses of obese mothers develop insulin resistance in utero. Diabetes Care. 2009 Jun;32(6):1076-80. doi: 10.2337/dc08-2077. PMID 19460915
- [Background] Mingrone G, Manco M, Mora ME, Guidone C, Iaconelli A, Gniuli D, Leccesi L, Chiellini C, Ghirlanda G. Influence of maternal obesity on insulin sensitivity and secretion in offspring. Diabetes Care. 2008 Sep;31(9):1872-6. doi: 10.2337/dc08-0432. Epub 2008 Jun 5. PMID 18535193
- [Background] Samuelsson AM, Matthews PA, Argenton M, Christie MR, McConnell JM, Jansen EH, Piersma AH, Ozanne SE, Twinn DF, Remacle C, Rowlerson A, Poston L, Taylor PD. Diet-induced obesity in female mice leads to offspring hyperphagia, adiposity, hypertension, and insulin resistance: a novel murine model of developmental programming. Hypertension. 2008 Feb;51(2):383-92. doi: 10.1161/HYPERTENSIONAHA.107.101477. Epub 2007 Dec 17. PMID 18086952
- [Background] Bayol SA, Simbi BH, Bertrand JA, Stickland NC. Offspring from mothers fed a 'junk food' diet in pregnancy and lactation exhibit exacerbated adiposity that is more pronounced in females. J Physiol. 2008 Jul 1;586(13):3219-30. doi: 10.1113/jphysiol.2008.153817. Epub 2008 May 8. PMID 18467362
- [Background] Muhlhausler BS, Duffield JA, McMillen IC. Increased maternal nutrition stimulates peroxisome proliferator activated receptor-gamma, adiponectin, and leptin messenger ribonucleic acid expression in adipose tissue before birth. Endocrinology. 2007 Feb;148(2):878-85. doi: 10.1210/en.2006-1115. Epub 2006 Oct 26. PMID 17068138
- [Background] Chang GQ, Gaysinskaya V, Karatayev O, Leibowitz SF. Maternal high-fat diet and fetal programming: increased proliferation of hypothalamic peptide-producing neurons that increase risk for overeating and obesity. J Neurosci. 2008 Nov 12;28(46):12107-19. doi: 10.1523/JNEUROSCI.2642-08.2008. PMID 19005075
- [Background] Walker CD, Naef L, d'Asti E, Long H, Xu Z, Moreau A, Azeddine B. Perinatal maternal fat intake affects metabolism and hippocampal function in the offspring: a potential role for leptin. Ann N Y Acad Sci. 2008 Nov;1144:189-202. doi: 10.1196/annals.1418.023. PMID 19076377
- [Background] Shankar K, Kang P, Harrell A, Zhong Y, Marecki JC, Ronis MJ, Badger TM. Maternal overweight programs insulin and adiponectin signaling in the offspring. Endocrinology. 2010 Jun;151(6):2577-89. doi: 10.1210/en.2010-0017. Epub 2010 Apr 6. PMID 20371699
- [Background] Aagaard-Tillery KM, Grove K, Bishop J, Ke X, Fu Q, McKnight R, Lane RH. Developmental origins of disease and determinants of chromatin structure: maternal diet modifies the primate fetal epigenome. J Mol Endocrinol. 2008 Aug;41(2):91-102. doi: 10.1677/JME-08-0025. Epub 2008 May 30. PMID 18515302
- [Background] Ng SF, Lin RC, Laybutt DR, Barres R, Owens JA, Morris MJ. Chronic high-fat diet in fathers programs beta-cell dysfunction in female rat offspring. Nature. 2010 Oct 21;467(7318):963-6. doi: 10.1038/nature09491. PMID 20962845
- [Background] Suter MA, Chen A, Burdine MS, Choudhury M, Harris RA, Lane RH, Friedman JE, Grove KL, Tackett AJ, Aagaard KM. A maternal high-fat diet modulates fetal SIRT1 histone and protein deacetylase activity in nonhuman primates. FASEB J. 2012 Dec;26(12):5106-14. doi: 10.1096/fj.12-212878. Epub 2012 Sep 14. PMID 22982377
- [Background] Sohi G, Marchand K, Revesz A, Arany E, Hardy DB. Maternal protein restriction elevates cholesterol in adult rat offspring due to repressive changes in histone modifications at the cholesterol 7alpha-hydroxylase promoter. Mol Endocrinol. 2011 May;25(5):785-98. doi: 10.1210/me.2010-0395. Epub 2011 Mar 3. PMID 21372147
- [Background] Gong L, Pan YX, Chen H. Gestational low protein diet in the rat mediates Igf2 gene expression in male offspring via altered hepatic DNA methylation. Epigenetics. 2010 Oct 1;5(7):619-26. doi: 10.4161/epi.5.7.12882. Epub 2010 Oct 1. PMID 20671425
- [Background] van Straten EM, Bloks VW, Huijkman NC, Baller JF, van Meer H, Lutjohann D, Kuipers F, Plosch T. The liver X-receptor gene promoter is hypermethylated in a mouse model of prenatal protein restriction. Am J Physiol Regul Integr Comp Physiol. 2010 Feb;298(2):R275-82. doi: 10.1152/ajpregu.00413.2009. Epub 2009 Nov 4. PMID 19889862
- [Background] Zheng S, Rollet M, Pan YX. Maternal protein restriction during pregnancy induces CCAAT/enhancer-binding protein (C/EBPbeta) expression through the regulation of histone modification at its promoter region in female offspring rat skeletal muscle. Epigenetics. 2011 Feb;6(2):161-70. doi: 10.4161/epi.6.2.13472. Epub 2011 Feb 1. PMID 20930553
- [Background] Zhou D, Pan YX. Gestational low protein diet selectively induces the amino acid response pathway target genes in the liver of offspring rats through transcription factor binding and histone modifications. Biochim Biophys Acta. 2011 Oct;1809(10):549-56. doi: 10.1016/j.bbagrm.2011.07.003. Epub 2011 Jul 18. PMID 21777709
- [Background] Jousse C, Parry L, Lambert-Langlais S, Maurin AC, Averous J, Bruhat A, Carraro V, Tost J, Letteron P, Chen P, Jockers R, Launay JM, Mallet J, Fafournoux P. Perinatal undernutrition affects the methylation and expression of the leptin gene in adults: implication for the understanding of metabolic syndrome. FASEB J. 2011 Sep;25(9):3271-8. doi: 10.1096/fj.11-181792. Epub 2011 Jun 13. PMID 21670064
- [Background] Zhang S, Rattanatray L, MacLaughlin SM, Cropley JE, Suter CM, Molloy L, Kleemann D, Walker SK, Muhlhausler BS, Morrison JL, McMillen IC. Periconceptional undernutrition in normal and overweight ewes leads to increased adrenal growth and epigenetic changes in adrenal IGF2/H19 gene in offspring. FASEB J. 2010 Aug;24(8):2772-82. doi: 10.1096/fj.09-154294. Epub 2010 Apr 6. PMID 20371620
- [Background] Raychaudhuri N, Raychaudhuri S, Thamotharan M, Devaskar SU. Histone code modifications repress glucose transporter 4 expression in the intrauterine growth-restricted offspring. J Biol Chem. 2008 May 16;283(20):13611-26. doi: 10.1074/jbc.M800128200. Epub 2008 Mar 7. PMID 18326493
- [Background] Vucetic Z, Kimmel J, Reyes TM. Chronic high-fat diet drives postnatal epigenetic regulation of mu-opioid receptor in the brain. Neuropsychopharmacology. 2011 May;36(6):1199-206. doi: 10.1038/npp.2011.4. Epub 2011 Feb 16. PMID 21326195
- [Background] Thompson RF, Fazzari MJ, Niu H, Barzilai N, Simmons RA, Greally JM. Experimental intrauterine growth restriction induces alterations in DNA methylation and gene expression in pancreatic islets of rats. J Biol Chem. 2010 May 14;285(20):15111-15118. doi: 10.1074/jbc.M109.095133. Epub 2010 Mar 1. PMID 20194508
- [Background] Tobi EW, Lumey LH, Talens RP, Kremer D, Putter H, Stein AD, Slagboom PE, Heijmans BT. DNA methylation differences after exposure to prenatal famine are common and timing- and sex-specific. Hum Mol Genet. 2009 Nov 1;18(21):4046-53. doi: 10.1093/hmg/ddp353. Epub 2009 Aug 4. PMID 19656776
- [Background] Durmus B, Arends LR, Ay L, Hokken-Koelega AC, Raat H, Hofman A, Steegers EA, Jaddoe VW. Parental anthropometrics, early growth and the risk of overweight in pre-school children: the Generation R Study. Pediatr Obes. 2013 Oct;8(5):339-50. doi: 10.1111/j.2047-6310.2012.00114.x. Epub 2012 Dec 13. PMID 23239588
- [Background] Drong AW, Lindgren CM, McCarthy MI. The genetic and epigenetic basis of type 2 diabetes and obesity. Clin Pharmacol Ther. 2012 Dec;92(6):707-15. doi: 10.1038/clpt.2012.149. Epub 2012 Oct 10. PMID 23047653
- [Background] Toperoff G, Aran D, Kark JD, Rosenberg M, Dubnikov T, Nissan B, Wainstein J, Friedlander Y, Levy-Lahad E, Glaser B, Hellman A. Genome-wide survey reveals predisposing diabetes type 2-related DNA methylation variations in human peripheral blood. Hum Mol Genet. 2012 Jan 15;21(2):371-83. doi: 10.1093/hmg/ddr472. Epub 2011 Oct 12. PMID 21994764
- See also: Florida Hospital Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org